CLINICAL TRIAL: NCT04931563
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Phase III Study Evaluating the Efficacy and Safety of Anifrolumab in Asian Participants With Active Systemic Lupus Erythematosus
Brief Title: Anifrolumab Asian PhIII Efficacy Study for Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3468C00003
Record Dates: First submitted 2021-04-29; First posted 2021-06-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Active Systemic Lupus Erythematosus
MeSH Terms: interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Placebo will be administered via controlled IV infusion pump into a peripheral vein over a minimum of 30 minutes Q4W from Week 0 to Week 48. Each dose must be at least 14 days apart.
  Interventions: Drug: placebo
- anifrolumab (Active Comparator): Anifrolumab will be administered via controlled IV infusion pump into a peripheral vein over a minimum of 30 minutes Q4W from Week 0 to Week 48. Each dose must be at least 14 days apart.
  Interventions: Biological: Anifrolumab

INTERVENTIONS:
Biological: Anifrolumab — Intravenous infusion (IV)
  Arms: anifrolumab
Drug: placebo — Intravenous infusion (IV)
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an intravenous treatment regimen of anifrolumab versus placebo in Asian participants with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase III, multicenter, multinational, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of an intravenous treatment regimen of 300 mg anifrolumab versus placebo in participants with moderate to severe, autoantibody positive SLE while receiving SOC treatment. The study will be performed in participants aged 18 to 70 years of age.

Participants with a confirmed diagnosis of moderate to severe active SLE and are currently receiving SOC comprising of oral corticosteroids (OCSs) and/or antimalarial, and/or immunosuppressants, either alone or any combination of them, for a required duration of treatment at a stable dose, as described in the inclusion criteria shall be included. Participants must have eligible scores for SLEDAI-2K, BILAG-2004, and PGA as confirmed by the DACRT.

Eligible participants will be randomised in a 1:1 ratio to receive either a fixed intravenous dose of 300 mg anifrolumab plus SOC or placebo plus SOC every 4 weeks (Q4W) for a total of 13 doses (Week 0 to Week 48), with the primary endpoint evaluated at the Week 52 visit.

ELIGIBILITY:
Key inclusion criteria:

1. Aged 18 to 70 years.
2. Body weight ≥ 40 kg.
3. Confirmed diagnosis of SLE(1997 ACR revised criteria) for ≥ 24 weeks.
4. Must be receiving at least one of the following SOC regimens at screening:

   1. oral prednisone monotherapy: ≥ 7.5 mg/day and ≤ 40 mg/day, stable for > 2 weeks;
   2. Immunosuppressant(s) with or without OCS and must be stable for ≥ 8 weeks;
   3. Oral prednisone plus immunosuppressant: start date, stability and maximum dose required.
5. At least one of these antibodies positive: ANA, anti-dsDNA and anti-Smith.
6. SLEDAI-2K score ≥ 6 points at screening and "Clinical" SLEDAI-2K score ≥4 points at both screening and Day1(randomisation), and BILAG with at least 1 level A organ system or 2 level B organ system, and PGA score ≥ 1.0 at screening.
7. Chest imaging shows no clinically significant abnormalities (unless due to SLE).
8. No evidence or medical history of active TB, indeterminate TB should be referred to a TB specialist.
9. All participants should use effective contraception methods as protocol requests.
10. Any negative SARS-CoV-2 RT-PCR test result at screening and no known or suspected COVID-19 infection or exposure within 2 weeks prior to screening and between screening and randomisation visits.

Key exclusion criteria:

1. History or current diagnose of clinically significant non-SLE related vasculitis, severe or unstable neuropsychiatric SLE, active severe SLE-driven renal disease, catastrophic anti-phospholipid syndrome, inflammatory joint or skin disease other than SLE, non-SLE disease that has required treatment of certain dosage of corticosteroid.
2. History or evidence of suicidal ideation or suicidal behavior.
3. History or current diagnose of MTCD or overlap syndrome, unless overlap with RA or MTCD which has developed into SLE.
4. History of recurrent infection requiring hospitalization and IV antibiotics, or opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years of randomization, or clinically significant chronic infection within 3 months, or recent infection still under treatment.
5. History of immunodeficient condition, HIV positive included.
6. Confirmed HBsAg positive, or HBcAb positive and HBV DNA detectable, or hepatitis C antibody positive.
7. History of severe case of herpes zoster.
8. Herpes zoster, CMV or EB infection which has not completely resolved within 12 weeks before screening.
9. Acute COVID-19 infection or history of severe COVID-19.
10. History of cancer, apart from cured squamous or basal cell carcinoma and cervical cancer in situ.
11. Female participants with abnormal pap smear results.
12. Prior receipt of anifrolumab ,or any commercially available Janus kinase (JAK) inhibitor ≤ 12 weeks or Bruton's tyrosine kinase (BTK) inhibitor ≤ 24weeks prior to signing the ICF; any investigational medicinal product(small molecule or biologic agent) within 4 weeks or 5 half-lives prior to signing of the ICF, whichever is greater.
13. Known history of allergy to any component of the IP formulation or protein related products.
14. Receipt of any of the following:

    1. Intramuscular or IV glucocorticosteroids within 6 weeks;
    2. Any live or attenuated vaccine within 8 weeks;
    3. Any restricted medication listed in protocol;
    4. Blood transfusion within 4 weeks. 15 Regular use of > 1 NSAID within 2 weeks or receipt of fluctuating doses of a NSAID within 2 weeks.

16. Certain laboratory test results requirements. 17. Concurrent enrolment in another clinical study. 18. History or current alcohol, drug or chemical abuse within 1 year. 19. Major surgery within 8 weeks or planned elective major surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of participants who are responders between anifrolumab and placebo | Week 52
  Composite endpoint (BICLA),a composite binary endpoint defined by meeting all of the following criteria:
  * Reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, where worsening is defined as ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B
  * No worsening from baseline in SLEDAI-2K, where worsening is defined as an increase from baseline of >0 points in SLEDAI-2K
  * No worsening from baseline in participants' lupus disease activity, where worsening is defined as an increase of ≥0.30 points on a 3-point PGA visual analogue scale (VAS)

SECONDARY OUTCOMES:
The proportion of participants who achieve SRI(4) response at week 52 | Week 52
  SRI(4) response defined by meeting all of the following criteria:
  * Reduction from baseline of ≥ 4 points in the SLEDAI-2K;
  * No new organ systems affected as defined by 1 or more BILAG-2004 A or 2 or more BILAG-2004 B items compared to baseline;
  * No worsening from baseline in the participants' lupus disease activity defined by an increase ≥0.30 points on a 3-point PGA VAS;
The proportion of participants who achieve an oral corticosteroid (OCS) dose ≤7.5 mg/day at Week 40, which is maintained through Week 52 in the subgroup of those with baseline OCS ≥10 mg/day | Week 52
  Maintained OCS reduction defined by meeting all of the following criteria:
  * Achieve an OCS dose of ≤7.5 mg/day prednisone or equivalent by Week 40
  * Maintain an OCS dose ≤7.5 mg/day prednisone or equivalent from Week 40 to Week 52
Annualized flare rate | Week 52
  Annualised flare rate with flare defined as either 1 or more new BILAG-2004 A or 2 or more new BILAG-2004 B items compared to the previous visit

CONTACTS AND LOCATIONS:
Locations (54):
- China (39):
  - Research Site, Baoding
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Binzhou
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chuangchun
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Jieyang
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xinxiang
  - Research Site, Yinchuan
  - Research Site, Zaozhuang
  - Research Site, Zhengzhou
- Research Site, Hong Kong, Hong Kong
- Philippines (5):
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Quezon City
- South Korea (3):
  - Research Site, Gwangju
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Research Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home